CLINICAL TRIAL: NCT03893188
Title: A Multicenter, Observational Cohort to Study the Characteristics of Individuals Asking for Pre-exposure Prophylaxis (PrEP) and the Incidence of HIV and Other Sexually Transmitted Infections: 'The SwissPrEPared Study'
Brief Title: The SwissPrEPared Study
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss HIV Cohort Study (Network); Federal Office of Public Health, Switzerland (Other Government); Positive Council Switzerland (Unknown); Cantonal Hospital of St. Gallen (Other); University Hospital, University of Bern (Unknown); Cantonal Hosptal, Baselland (Other); University Hospital, Geneva (Other); University of Lausanne Hospitals (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC-Nr.2018-02015
Record Dates: First submitted 2019-03-14; First posted 2019-03-28 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: HIV Preexposure Prophylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People asking for PrEP: All individuals aged >18 years asking for PrEP prescription at one of the participating centers will be asked to participate to the SwissPrEPared Study(consecutive ongoing recruitment). Only HIV negative individuals will be deemed eligible.

SUMMARY:
Nested within the SwissPrEPared Program, the "SwissPrEPared Study" - a large, multicentric, nation-wide cohort study - aims to longitudinally follow individuals asking for PrEP prescription over a period of 3 years.

DETAILED DESCRIPTION:
The main aims of the study will be:

1. To obtain epidemiological data on individuals asking for PrEP in Switzerland. We are particularly interested in:

   * Determining the extent of PrEP use in Switzerland;
   * Assessing and monitoring the occurrence of sexually transmitted infections (STIs) in this particular population.
2. To assess sexual health and sexual well-being in individuals asking for PrEP using a questionnaire specifically designed for the SwissPrEPared program.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the SwissPrEPared program
* Aged ≥16 years
* HIV negative

Exclusion Criteria:

* Individuals unable to follow program procedures (e.g. language barriers, mental or psychiatric disorders)

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals aged >16 years asking for PrEP prescription at one of the participating centers will be asked to participate to the SwissPrEPared study (consecutive ongoing recruitment). Only HIVnegative individuals will be deemed eligible. Participants for whom PrEP is not indicated or individuals declining PrEP will still be offered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Number of individuals asking for PrEP | 10 years
  Number of individuals asking for PrEP
Proportion of individuals qualifying for PrEP according to current guidelines | 10 years
  Proportion of individuals qualifying for PrEP according to current guidelines
PrEP regime used (daily, intermittent, on-demand) | 10 years
  PrEP regime used (daily, intermittent, on-demand)
Mode of drug supply (pharmacy versus online) | 10 years
  Mode of drug supply (pharmacy versus online)
Adherence rates to programme | 10 years
  Adherence rates to programme assessed via lost to follow-up and dropouts
Adherence rates to PrEP | 10 years
  Adherence rates to PrEP measured via self-report questionnaire
Occurrence of side effects | 10 years
  Occurrence of side effects
Prevalence of HIV | 10 years
  Prevalence of HIV
Incidence of HIV | 10 years
  Incidence of HIV
Prevalence of other STIs (syphilis, hepatitis B, hepatitis C, gonorrhoea, chlamydia, mycoplasma genitalium) | 10 years
  Prevalence of other STIs (syphilis, hepatitis B, hepatitis C, gonorrhoea, chlamydia, mycoplasma genitalium)
Incidence of other STIs (syphilis, hepatitis B, hepatitis C, gonorrhoea, chlamydia, mycoplasma genitalium) | 10 years
  Incidence of other STIs (syphilis, hepatitis B, hepatitis C, gonorrhoea, chlamydia, mycoplasma genitalium)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hampel, MD, Principal Investigator — University of Zurich
Locations (41):
- Switzerland (41):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Kantonsspital Baden, Baden, Canton of Aargau
  - MedCenter Volta, Basel, Canton of Basel-City
  - Praxis Hammer, Basel, Canton of Basel-City
  - Praxis dr. med. Clara Thierfelder, Basel, Canton of Basel-City
  - University Hospital Basel, Basel, Canton of Basel-City
  - Spitalzentrum Biel - Centre hospitalier Bienne, Biel/Bienne, Canton of Bern
  - Spital Thun, Thun, Canton of Bern
  - Médecine Interne/Infectiologie FMH, Cottens, Canton of Fribourg
  - Hôpital du Jura, Delémont, Canton of Jura
  - Kantonsspital Olten, Olten, Canton of Solothurn
  - Medical and Therapeutic Centre La Lignière, Gland, Canton of Vaud
  - Cabinet Dr. Erika Castro Batänjer, Lausanne, Canton of Vaud
  - Cabinet Gare 10, Lausanne, Canton of Vaud
  - Cabinet Rumine 35, Lausanne, Canton of Vaud
  - Cabinet Rumine 9, Lausanne, Canton of Vaud
  - University Hospital Laussane, Lausanne, Canton of Vaud
  - Checkpoint Lausanne, Lausanne, Canton of Vaud
  - Fondation PROFA, Renens VD, Canton of Vaud
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - Kantonsspital Münsterlingen, Münsterlingen, Thurgau
  - Kantonsspital Ticcino, Lugano, Ticcino
  - Checkpoint Bern, Bern
  - University Hospital Bern, Bern
  - Cabinet Dr. Marta Buzzi, Geneva
  - Praxis Emmanuelle Boffi, Geneva
  - University Hospital Geneva, Geneva
  - Cabinet Malagnou 2, Geneva
  - Checkpoint Geneva, Geneva
  - Maihofpraxis, Lucerne
  - Réseau Hospitalier Neuchâtelois, Neuchâtel
  - Kantonspital St. Gallen, Sankt Gallen
  - ARUD, Zurich
  - Travel Clinic UZH, Zurich
  - Praxis Kalkbreite, Zurich
  - Checkpoint Zürich, Zurich
  - Dermatologisches Zentrum Zürich AG, Zurich
  - Praxisgemeinschaft D29, Zurich
  - Stadtspital Triemli, Zurich
  - Division of Infectious Diseases and Hospital Epidemiology, University Hospital Zurich, University of Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the study protocol (including the statistical plan) will be available after de-identification of participants following article publication. Data will be provided to investigators whose proposed use of the data has been approved by the study team and the Scientific Board of the Swiss HIV Cohort Study. Proposals should be directed to jan.fehr@usz.ch.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Hovaguimian F, Martin E, Reinacher M, Rasi M, Schmidt AJ, Bernasconi E, Boffi El Amari E, Braun DL, Calmy A, Darling K, Christinet V, Depmeier C, Hauser C, Lauchli S, Notter J, Stoeckle M, Surial B, Vernazza P, Bruggmann P, Tarr P, Haerry D, Bize R, Low N, Lehner A, Boni J, Kouyos RD, Fehr JS, Hampel B. Participation, retention and uptake in a multicentre pre-exposure prophylaxis cohort using online, smartphone-compatible data collection. HIV Med. 2022 Feb;23(2):146-158. doi: 10.1111/hiv.13175. Epub 2021 Oct 3. PMID 34605153

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03893188/Prot_SAP_000.pdf